CLINICAL TRIAL: NCT05605457
Title: Clinical Performance of Nanohybrid Resin Composite Lined With PRG Barrier Coat Compared to Resin Modified Glass Ionomer in Class V Carious Cavities Over 18 Months: Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nora Ahmed Salah, assistant lecturer at Badr University in Cairo, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRG barrier coat liner Class V
Record Dates: First submitted 2022-10-29; First posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Class V Dental Caries
Keywords: PRG barrier coat; nanohybrid resin composite; Resin modified glass ionomer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- PRG barrier coat (Experimental): It is a light cured surface-partially reacted glass (S-PRG) filler particles with a multifunctional glass core embedded in a resin matrix.
  Interventions: Device: PRG barrier coat + nanohybrid composite
- Resin modified glass ionomer (Active Comparator): Resin modified glass ionomer (Fuji II LC, GC, Japan). RMGIC are glass-ionomer cements with small quantity of monomers and initiators so the acid-base reaction is supplemented by a second polymerization reaction.
  Interventions: Device: resin modified glass ionomer

INTERVENTIONS:
Device: PRG barrier coat + nanohybrid composite — It is a light cured surface-partially reacted glass (S-PRG) filler particles with a multifunctional glass core embedded in a resin matrix.
  Arms: PRG barrier coat
Device: resin modified glass ionomer — RMGIC are glass-ionomer cements with small quantity of monomers and initiators so the acid-base reaction is supplemented by a second polymerization reaction
  Arms: Resin modified glass ionomer

SUMMARY:
Class V carious lesions will be restored using two different restorative materials either Resin modified glass ionomer or nanohybrid resin composite lined by PRG barrier coat. Each restoration will be evaluated for clinical parameters after finishing and polishing at baseline, at 6 months, 12 months and at 18 months. The restorations will be clinically examined according to modified USPHS criteria in terms of retention, marginal adaptation, marginal discoloration, secondary caries and postoperative sensitivity.

DETAILED DESCRIPTION:
Class V carious lesions will be restored using two different restorative materials either resin modified glass ionomer or nanohybrid resin composite lined by PRG barrier coat.Each restoration will be evaluated for clinical parameters after finishing and polishing at baseline, at 3 months, 6 months, 12 months and at 18 months. The restorations will be clinically examined according to modified USPHS criteria in terms of retention, marginal adaptation, marginal discoloration, secondary caries and postoperative sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years Males or females. Patients with untreated cervical carious lesion that need restoration. Participants available for recall Patients with moderate to high caries risk

Teeth Inclusion Criteria No spontaneous pain Absence of tooth mobility

Exclusion Criteria:

* Patients with para-functional habits Experience with allergic reactions against any component of used materials. Teeth Exclusion Criteria Non-vital teeth Teeth with orthodontic appliance Teeth with advanced periodontal diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Modified USPHS criteria | 18 months
  Retention, marginal discoloration, marginal adaptation, secondary caries

SECONDARY OUTCOMES:
Modified USPHS criteria | 18 months
  Postoperative hypersensitivity